CLINICAL TRIAL: NCT06230003
Title: Efficacy of Erector Spinae Plane (ESP) Block in Patients With Inflammatory Bowel Disease (IBD) Undergoing Major Abdominal Surgery: A Double-Blind Randomized Control Trial
Brief Title: Efficacy of Erector Spinae Plane (ESP) Block in Patients With Inflammatory Bowel Disease (IBD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Principal Investigator, Dr. Naveed Siddiqui, Associate Professor, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-0272-A
Record Dates: First submitted 2023-11-24; First posted 2024-01-29 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2024-02

CONDITIONS: Opioid Use
MeSH Terms: interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): Ultrasound guided bilateral ESP block either with local anesthetic
  Interventions: Drug: Ropivacaine
- Control group (Placebo Comparator): Ultrasound guided bilateral ESP block either with normal saline
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Ropivacaine — Ultrasound guided ESP block either with the local anesthetic of 0.5% of Ropivicane 20 mL bilaterally (intervention group) or normal saline (control group) before surgery which will take 5-10 minutes in a 1:1 ratio.
  Arms: Intervention group
Drug: normal saline — Ultrasound guided bilateral ESP block either with normal saline
  Arms: Control group

SUMMARY:
This will be a prospective, double-blind randomized controlled clinical trial. There will be two arms of treatment: intervention and control group. Preoperatively patients will be allocated at random to receive ultrasound guided bilateral ESP block either with the local anesthetic (intervention group) normal saline (control group). The aim of this study is to examine the effect of ESP block to increase the Quality of Recovery (measured via QoR-15 total score) and decrease opioid consumption.

DETAILED DESCRIPTION:
Work Plan: This prospective trial would include Inflammatory Bowel Disease (IBD) patients undergoing laparoscopic or laparoscopic assisted abdominal surgery. Patients generally have pre-anesthetic visits 1-2 weeks prior to their scheduled operation. Patients identified by the clinical Research Study Assistant (CRSA) based on inclusion and exclusion criteria, will be approached regarding this study in the pre-anesthetic clinic. Patients will be made aware of the components of the study and the CRSA will be present to answer any questions. Patients will be allocated at random to receive ultrasound guided (Erector spinae plane) ESP block either with the local anesthetic of 0.5% of Ropivicane 20 mL bilaterally (intervention group) or normal saline (control group) before surgery which will take 5-10 minutes in a 1:1 ratio. Anesthesiologist and patients will be blinded of the allocation. Allocation sequence will be concealed using opaque, sealed, consecutively numbered envelopes. Written informed consent will be obtained from all participants after confirmation of eligibility. Baseline measurements will be made by the CRSA in the pre-anesthetic Clinic. The study coordinator will collect the data once a day for maximum 10 minutes each time up to 3 days postoperatively. There will be a virtual (via telephone) follow up data for quality of life (QoL) at "6 weeks" post-discharge. Sample Size: Sample size justification was based on the primary outcome, QoR15, and the primary objective. According to the previous report10 and our preliminary data, the mean (std) of the total score of QoR15 (quality of recovery) was conservatively assumed as 98 for patients in control group. The investigators estimated a sample size of 84 (42 per group) will achieve 80% power to detect an absolute 10 point increase in total score of QoR15 for patients in intervention group compared to the control group. A two-sided two-sample equal-variance t-test was used for the power analysis assuming a significance level of 0.05. To account for possible 5% lost follow up, the investigators will recruit a total of 90 patients for this study.

Performance of ESP block: Patient Selection. A thorough history, physical exam, and informed consent are carried out. Altered mental status, concomitant injuries, and intubation/ ventilation are considerations primarily with regard to the ability to position the patient safely and access the Paraspinal area to perform the block. The investigators do not view coagulopathy or the use of anticoagulants or antiplatelet drugs as absolute contraindications to ESP block because the theoretical risk of clinically significant hemorrhage or hematoma is very low; however, an individualized risk-benefit assessment should be performed for every patient. Block Equipment and Preparation. In the majority of patients, the investigators will use a high-frequency (10-15 MHz) linear-array transducer because it provides a higher-resolution image; however, a low-frequency (5-2 MHz) curvilinear probe is useful in more obese patients where the transverse processes lie at a depth greater than 4 cm. The block is performed before induction of anesthesia with full aseptic precautions, and the usual precautions for any regional anesthesia procedures will be applied. Scanning Technique. After patients are positioned optimally (sitting or lateral decubitus), the affected area is identified along with the target transverse process. The ultrasound transducer is placed in a longitudinal parasagittal orientation, about 3 cm lateral to the spinous processes, allowing for visualization of adjacent transverse processes (TP) in an in-plane approach. These are recognizable as flat, squared-off acoustic shadows with only a very faint image of the pleura visible. After correct TP identification, an 22-gauge echogenic needle (Pajunk E-Cath, Pajunk Medical Systems) is inserted using an in-plane, cranial-to-caudal approach to contact the bony shadow of the TP with the tip deep to the fascial plane of the erector spinae muscle. The correct location of the needle tip is confirmed by injecting 0.5-1 ml of normal saline 0.9% and observing linear fluid spread lifting the erector spinae muscle off the tip of the TP. Once the fascial plane is recognized, 20 mL of ropivacaine 0.5% is injected and cranial and caudal spread of local anesthetic can be visualized.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18-85 years old) diagnosed with IBD
2. ASA physical status I-III
3. IBD abdominal laparoscopic assisted surgeries under general anesthesia

Exclusion Criteria:

1. Unable to communicate in English
2. Unstable requiring emergency surgery
3. Open laparotomies
4. Morbidly obese
5. Pregnant
6. On chronic opioid treatment
7. Known allergies to local anesthetics
8. Altered mental status
9. Concomitant injuries.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery (via QoR-15) total score | baseline, 24 hours, 48 hours and 72 hours postoperatively
  This will be measured via QoR-15 (Quality of Recovery-15 questionnaire) where, "0" means the worst and "15" the best outcome.

SECONDARY OUTCOMES:
The intensity of postoperative pain | baseline, 24 hours, 48 hours and 72 hours postoperatively
  Pain will be measured by Visual Analog Scale (VAS) at rest and movement once a day using categorical pain scoring system. The scores are from 1 to 10, in which, 10 is the worse pain.
Opioid consumption | 24 hours, 48 hours and 72 hours postoperatively
  Total opioid consumption will be measured as 24-hour PCA usage each day up to 3 days postoperatively
Opioid related side effects | baseline, 24 hours, 48 hours and 72 hours postoperatively
  The side effects of opioids will be measured using Opioid-related symptom Distress Scale (ORSDS). The answers to each side effects will be either "ye" or "no".
The hospital LOS | From admission to the hospital until discharge, an average of 5 days
  The hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Siddiqui, MD, Principal Investigator — Associate Professor
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No